CLINICAL TRIAL: NCT03446235
Title: Feasibility and Explorative Study to Test the Superiority of Connected Health Care Using Wearable Device to Improve Body Composition and Fitness Level
Brief Title: Connected Health Care in Exercise Program for Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Regis Fernandes, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-004529
Record Dates: First submitted 2018-01-11; First posted 2018-02-26 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Physical Activity; Exercise
Keywords: Obesity; Physical Activity; Exercise; Wearable device
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Motivational Interviewing; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected Health (Experimental): This group will get 2 interviews about physical exercise (exercise instruction with motivational interview) and 6 communications with individualized instruction and counseling of their physical exercise (investigators can access activity data and exercise log) including the usage of the monitoring device.
  Interventions: Behavioral: Exercise instruction with motivational interview
- Self-Monitoring (Active Comparator): This group will do physical exercise following the initial instruction and self-monitor them. Investigators can access activity data and exercise log but will not discuss with the subjects about the data.
  Interventions: Behavioral: Self-monitoring

INTERVENTIONS:
Behavioral: Exercise instruction with motivational interview — An activity tracker and a heart rate monitor to track the participants activity and exercise records will be used. In addition to the basic instruction of exercise and nutrition, an exercise physiologist provides individualized exercise instruction with a motivational interviewing skill, which is a different style from traditional persuasive style of communication between the healthcare professionals and patients.
  Arms: Connected Health
Behavioral: Self-monitoring — An activity tracker and a heart rate monitor to track the participants activity and exercise records will be used. Basic instruction about exercise and nutrition is provided at the initial visit.
  Arms: Self-Monitoring

SUMMARY:
Many kinds of wearable technology have become available, but the superiority of those devices in weight loss compared to the standard care without them is uncertain. The possible problems are long-term self-motivation, utility and validity of the device, and outcome measures in clinical trials. The connected health care with motivational interviewing as an intervention, and body composition parameters in addition to body weight as outcome measures are employed in the project. The expected outcome is that connected health care, which is more individualized approach by heath care professionals, is more effective compared to self-monitoring using wearable devices. Two types of wearable device are going to be used to monitor 1) body activity and 2) heart rate variables during exercise which reflect fitness level in this study in order to investigate appropriate monitoring parameters to predict outcome measures.

The hypothesis is that addition of connected health system will result in improvement of body composition and fitness level compared to self-monitoring.

DETAILED DESCRIPTION:
Patients with age 18 to 59 years old and body mass index between 30 to 39.9 are to be enrolled at Mayo Clinic in Arizona. All enrolled subjects receive wearable monitoring devices with remote tracking capability and brochure regarding nutrition and physical exercise with basic instruction. Subjects are randomly assigned to connected health care group versus self-monitoring group. Connected health care group will have 2 interviews about physical exercise and 6 communications with individualized instruction and counseling of their exercise including the usage of the monitoring devices. Self-monitoring group will do physical exercise following the initial basic instruction and self-monitor them.

All subjects visit Mayo Clinic to get outcome measures at 0, 12, and 24weeks. Outcome measures will be compared before, at 12 weeks, and after the 24 weeks of the fitness program.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index of 30 to <40 kg/m^2

Exclusion Criteria:

* End of organ damage from hypertension
* Diabetes
* Liver disease
* Chronic lung disease
* Neuromuscular disease
* Any conditions that limit exercise
* Currently involved in other weight program

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Waist circumference | Baseline and 24 weeks
  Waist circumference is measured by tape at the end expiration while the patient is standing. Units centimeters.

SECONDARY OUTCOMES:
Change in weight | Baseline and 24 weeks
  Weight is measured using a commercially available body weight scale (TANITA body composition monitors). Units kg.
Change in body fat percentage | Baseline and 24 weeks
  Body fat percentage is measured using a commercially available body fat scale (TANITA body composition monitors). Units percentage.
Change in physical activity score | Baseline and 24 weeks
  International Physical Activity Questionnaire is filled out by patients. The International Physical Activity Questionnaire Long Form (IPAQ) (www.ipaq.ki.se) is to assess levels and patterns of physical activity.
  Continuous score expressed as "MET (metabolic equivalent)-min/week: MET level*minutes of activity/day*days per week" is calculated. Higher number means higher level of physical activity that a subject performed during last 7 days. The estimated range is from 0 to 3000. Units MET-minutes.
Change in Physical Activity Vital Sign | Baseline and 24 weeks
  Physical Activity Vital Sign (PAVS) (Greenwood JL, 2010) is a short physical activity assessment using closed ended questions to ask how many days a subject performed physical activity during the past week. Higher number means a subject spent more days on performing physical activity.
  The range is from 0 to 7. Units days.
Change in Veterans Specific Activity Questionnaire | Baseline and 24 weeks
  Veterans Specific Activity Questionnaire (VASQ) (Myers J, 2001) is a brief self administered questionnaire to predict exercise capacity (METs, metabolic equivalents). A subject select the minimum activity level that cause fatigue, short of breath, or discomfort. Higher number means higher fitness level of a subject. the range is from 1 to 13. Units METs.
Change in heart rate variables | Baseline and 24 weeks
  Heart rate recovery after 6 minute walk test is evaluated. Units beats/minute.
Change in 6 minute walk test | Baseline and 24 weeks
  Walking distance is evaluated. Units meters.

CONTACTS AND LOCATIONS:
Overall Officials: Regis I Fernandes, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States